CLINICAL TRIAL: NCT03368560
Title: A Breathing-Based Meditation Intervention for Patients With Treatment-Resistant Late Life Depression (TR-LLD): A Phase II Trial and Feasibility Study
Brief Title: A Breathing-Based Meditation Intervention for Patients With Treatment Resistant Late Life Depression
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding was not received.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Akshya Vasudev, MBBS, MD, MRCPsych, PG Cert Medical Education Associate Professor of Psychiatry and Medicine, Western University Consultant Geriatric Psychiatrist, London Health Sciences Centre, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110791
Record Dates: First submitted 2017-11-27; First posted 2017-12-11 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Late Life Depression
Keywords: Treatment-resistant Late Life Depression; Sudarshan Kriya Yoga; Glutathione

STUDY DESIGN:
Intervention Model Description: This study will recruit 30 patients with treatment-resistant late life depression, and 7 age-matched controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sudarshan Kriya Yoga (Active Comparator): Thirty participants with treatment-resistant late life depression (TR-LLD) will attend 5 instructional days of Sudarshan Kriya Yoga (SKY), followed by 3 weekly follow-ups, and 8 weeks of bimonthly follow-ups. Participants will also practice SKY for 25 minutes per day at home. These participants will attend 4 mental health assessments at weeks 0, 4, 8, and 12. Thirteen of the recruited TR-LLD will attend an MRI at baseline and post-intervention.
  Interventions: Other: Sudarshan Kriya Yoga
- Control (No Intervention): The seven recruited age-matched controls will complete a screening appointment and an MRI only for comparison. Demographic information will also be collected from the control participants. These individuals will not undergo the study intervention.

INTERVENTIONS:
Other: Sudarshan Kriya Yoga — Sudarshan Kriya Yoga (SKY): A 12-week training course conducted by certified instructors from the Art of Living Foundation. SKY training will take place in group-format (group sizes of 8-15 participants) in an appropriately sized and accessible community hall in London, Ontario.SKY training involves attending a week-long (5 days) course that teaches the basic principles of SKY over 2.5-3 hour daily sessions. This will be followed by once weekly follow up sessions (90 min/wk) for 3 weeks and then bimonthly sessions (every 2 weeks) for the next 8 weeks. In addition, participants will be asked to practice SKY at home daily (25 min/day) throughout the duration of the study period and log practice frequency and any other noteworthy observations in a log sheet that will be provided to them . Nutritional snacks will be provided during the 5 day SKY training course.
  Arms: Sudarshan Kriya Yoga

SUMMARY:
Late-life depression affects 2-8% of seniors and causes high rates of caregiver distress and risk of suicide. To exacerbate the problem, antidepressants, the cornerstone of therapy, are resistant in 55-80% of this population. Hence, this group of patients is labeled as having treatment-resistant late-life depression (TR-LLD).

Non-pharmacological interventions like meditation could offer significant benefits as augmentation strategies to improve response rate of antidepressants in TR-LLD. One such breath-based meditation intervention called Sudarshan Kriya Yoga is of interest based on highly significant preliminary data in adult patients with treatment-resistant depression, its scalability and relatively low cost to learn this lifelong skill.

Thirty patients diagnosed with TR-LLD will learn this intervention over 5 consecutive days by a certified para-professional trainer. This will be followed by 3 weekly 90 min follow-up sessions and then bimonthly sessions for 8 more weeks. SKY consists of a series of breathing techniques, including Sudarshan Kriya (SK), a sequential rhythm-specific breathing exercise. Participants will be asked to practice this technique for 25-30 minutes daily over the next 11 weeks. The investigators will collect clinical as well as feasibility outcome measures. The investigators will also explore if it is feasible to assess the antioxidant Glutathione (GSH) in the brain using a sophisticated magnetic resonance spectroscopy. The investigators suspect that GSH levels are reduced in TR-LLD and they will improve with SKY.

DETAILED DESCRIPTION:
RECRUITMENT AND CONSENT:

Patients will be recruited from Victoria Hospital, London Health Sciences Centre or Parkwood Mental Health, St. Joseph's Health Care London. Patients will be screened and recruited after giving valid consent.

STUDY INTERVENTION (Sudarshan Kriya Yoga, SKY):

The 30 recruited TR-LLD participants will be invited to attend training sessions on SKY. The SKY program is a highly structured and standardized mind-body resilience building program. Through SKY breathing, interactive discussions, journaling, yoga and guided meditations, the workshop builds a framework for resilience and empowerment, and develops self-awareness, connectedness and community, and a positive outlook. This is a minimally invasive treatment and is not routinely available as standard of care. SKY involves rhythmic, cyclical forms of breathing in which there are no pauses between inhalation and exhalation. The breathing practices of this program include: (a) a three-stage Pranayama with Ujjayi, also called Victory Breath or Ocean Breath (b) Bhastrika or Bellow's Breath and (c) Sudarshan Kriya (SK) or the Rhythmic Breath Technique.

SKY will be consistently taught to the participants by two instructors from The Art of Living Foundation, an international humanitarian and charitable organization. SKY training will take place in a group-format with group sizes varying between 4-6 participants. The investigators will conduct these training sessions in an appropriately sized and accessible community hall in London, Ontario. SKY training involves attending a 5-day course that teaches the basic principles of SKY over 2.5-3 hour daily sessions. These will be followed by once weekly follow up sessions (90 min/wk) for 3 weeks and then bimonthly sessions (every 2 weeks) for the next 8 weeks. In addition, participants will be asked to practice SKY at home daily (25 min/day) throughout the duration of the study period and log practice frequency and any other noteworthy observations in a log sheet that will be provided to them.

MENTAL HEALTH ASSESSMENTS:

Participants will be screened for eligibility using criteria described below , the Anti-Depressant Treatment History Form, and if applicable an MRI pre-screening checklist. Prior to the start of the intervention, trained raters will meet with eligible participants to obtain demographic information. Participants will complete baseline measures of depression, comorbid anxiety, quality of life and caregiver burden. Specifically, the following scales will be administered: Hamilton Depression Rating Scale (HAM-D 17 item version), Geriatric Anxiety Inventory, European Quality of Life (EQ-5D-5L) and the Zaritz Caregiver burden. The abovementioned scales will be administered again at three other time points, weeks 4, 8 and 12.

MRI:

Seven healthy control participants will be recruited by advertising via flyers in waiting areas of the clinic. In addition, spouses and other family members accompanying the patient, who appear to be of eligible age, will be offered a letter of information about this research study. All thirty recruited TR-LLD participants will also be offered the option of participating in the MRI portion of the study in addition to the study activities described above. Our goal is to recruit 13 TR-LLD to complete MRI scans.

All MRI participants will complete the MRI screening questionnaire. Control participants will additionally be asked to complete a Mini Neuropsychiatric Interview (MINI) to confirm an absence of any mental health diagnosis. Both control and TR-LLD participants who are eligible to take part in the MRI portion of the study will be asked to attend a one-hour appointment at the Western Centre for Functional and Metabolic Mapping at University Hospital campus of LHSC. Control participants will attend only one such appointment, while TR-LLD participants will be asked to attend one MRI visit pre-intervention and one MRI visit post-intervention. The Research Coordinator or Research Assistant will accompany participants to the MRI visit, while the MRI analysis itself will be completed by an in-house MRI technician at the Western Centre for Functional and Metabolic Mapping.

The investigators will conduct semi-structured interviews by trained raters on study completers as well as drop outs. If a participant consented to be part of the study but then decided against participation at any point, he/she will be offered the opportunity to identify any problems with our approach by participating in a short interview conducted by a trained research assistant.

ELIGIBILITY:
Inclusion Criteria:

* 60-80 years of age
* major depressive disorder, as per the results of an interview by a trained rater using the Structured Clinical Interview for DSM-5 and subsequently confirmed by the psychiatrist
* Mild to moderate depression as confirmed by a score on the HAM-D 17 between 8 and 23
* Have failed at least two trials of antidepressants, given at adequate doses for adequate duration during the current episode
* Able to follow verbal instructions and sit without physical discomfort for 45 minutes
* Willing and able to attend at least 75% of all Sudarshan Kriya Yoga (SKY) sessions
* Willing to dedicate 25-30 minutes/day to SKY practice at home
* Low risk of suicide based on a clinical initial interview and during follow-up interviews at weeks 4, 8 and 12.

Exclusion Criteria:

* Uncontrolled hypertension, seizure disorder, psychosis, substance abuse, or dementia
* Currently participating in other similar studies or currently practicing any type of formal meditation, mindfulness or breathing techniques
* A major surgery within 6 weeks prior to commencement of or scheduled during, the study intervention
* A traumatic brain injury
* Any contraindications to MRI will also be excluded
* Healthy control participants must have no significant mental health issues, or contraindications to MRI.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Severity of TR-LLD as measured by the Hamilton Depression Scale (HAM-D17). | 12 weeks
  The primary outcome measure will be the Hamilton Depression Rating Scale (HAM-D 17) score. The HAM-D17 rates symptoms commonly associated with Major Depressive Disorder (MDD). A total score is calculated based on the first 17 questions of the HAM-D with a score range of 0 to 53. A higher score indicates more severe depression, and a lower score indicates fewer and/or less severe symptoms of depression.

SECONDARY OUTCOMES:
Glutathione levels measured by a 7-Tesla Magnetic Resonance Imaging (7T-MRI) in TR-LLD. | 12 weeks
  Brain glutathione (GSH) levels, a measure of inflammatory stress, will be measured in the prefrontal cortex at baseline and after 12-weeks of SKY intervention via sophisticated magnetic resonance spectroscopy for TR-LLD. Control participants will complete one such measurement.
Caregiver burden in caregivers of TR-LLD as measured by the Zaritz Caregiver Burden scale. | 12 weeks
  The Zaritz Caregiver Burden scale will be administered to caregivers of TR-LLD participants. This scale indicates the burden placed on caregivers by providing care for TR-LLD patients. A total score will be calculated, with scores ranging from 0 to 88. A lower score indicates little to no burden while a higher score indicates severe burden.
Quality of Life of TR-LLD participants using the European Quality of Life (EQ-5D-5L) scale. | 12 weeks
  The European Quality of Life (EQ-5D-5L) scale will be used to assess the quality of life of study participants. This scale has two scores; the descriptive system and the EQ Visual Analogue scale (EQ VAS). The descriptive system consists of 5 questions each with 5 possible answers allowing for 5 possible health states. A score of 1 indicates no problems with the 5 measured dimensions, while a score of 5 would indicate the most severe possible state for each dimension. The descriptive system includes 5 sub-scores ranging from 1 (no issues) to 5 (severe problems), which will be converted to a specific single index value. The EQ VAS consists of only one question ranging from 0 (worst possible state of health) to 100 (best possible state of health).
Anxiety severity of TR-LLD participants measured by the Geriatric Anxiety Inventory (GAI). | 12 weeks.
  The Geriatric Anxiety Inventory (GAI) assesses anxiety in geriatric patients. The questionnaire consists of 20 agree or disagree questions with total scores ranging from 0 (no anxiety) to 20 (severe anxiety).

IPD SHARING:
Plan to Share IPD: No